CLINICAL TRIAL: NCT07067125
Title: A Qualitative Evaluation of the Effects of Augmented Reality-Supported Training Methods on Body Awareness and Exercise Adherence in Adolescents With Idiopathic Scoliosis
Brief Title: Augmented Reality-Assisted Physiotherapy for Adolescents With Idiopathic Scoliosis: A Qualitative Study
Acronym: AR-AIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Merve Karatel, Assistant Professor, Hasan Kalyoncu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/060; 323s271 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye (TÜBİTAK))
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Scoliosis Idiopathic Adolescent; Scoliosis Idiopathic Adolescent Treatment
Keywords: Adolescent idiopathic scoliosis; augmented reality; qualitative research; psychosocial adjustment; physiotherapy

STUDY DESIGN:
Intervention Model Description: This study utilizes a single-group interventional design in which all participants will receive augmented reality-supported physiotherapeutic scoliosis-specific exercises for a minimum of four weeks. The intervention will be delivered by licensed physiotherapists using a standardized protocol that includes real-time visual feedback and interactive training components. No control or comparison group is included. This design was selected to qualitatively explore participants' individual experiences, perceptions of body awareness, motivational responses, and adherence behaviors during AR-based rehabilitation. Data will be collected through post-intervention interviews.
Masking Description: This is an open-label single-group study; no parties will be masked during the intervention or data collection processes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AR-Supported Physiotherapy Group (Experimental): Adolescents in this arm will receive scoliosis-specific physiotherapy supported by AR for a minimum of four weeks. The intervention includes real-time avatar feedback, interactive postural training, and gamified components. Exercises are delivered by licensed physiotherapists using a standardized AR interface. This group is designed to evaluate participants' experiences of body awareness, motivation, and adherence in technology-integrated conservative scoliosis care.
  Interventions: Behavioral: AR-Supported Scoliosis-Specific Physiotherapy

INTERVENTIONS:
Behavioral: AR-Supported Scoliosis-Specific Physiotherapy — This intervention consists of scoliosis-specific physiotherapy supported by AR technology. Participants will engage in postural correction exercises delivered by licensed physiotherapists using an AR system that provides real-time avatar feedback, movement guidance, and gamified motivation. The intervention aims to improve body awareness, adherence, and motivation among adolescents diagnosed with AIS. Each participant will complete at least four weeks of structured AR-supported sessions.
  Other Names: AR-Physio

SUMMARY:
This study aims to explore the effects of augmented reality (AR)-supported physiotherapy on body awareness, motivation, and exercise adherence in adolescents diagnosed with Adolescent Idiopathic Scoliosis (AIS). Using a qualitative phenomenological approach, the study will involve semi-structured interviews with adolescents who have completed at least four weeks of AR-based physiotherapeutic scoliosis-specific exercises. The goal is to understand participants' lived experiences with AR-enhanced rehabilitation and to inform the development of adolescent-centered, technology-integrated physiotherapy strategies in conservative scoliosis care.

DETAILED DESCRIPTION:
This prospective qualitative study is designed to examine how adolescents with AIS experience AR supported physiotherapeutic scoliosis-specific exercises. A phenomenological design was selected to capture participants' lived experiences, perceptions of body awareness, and motivational responses to the intervention. The study will be conducted in a physiotherapy unit in Türkiye, with ethics approval obtained from the institutional review board. Eligible participants will include adolescents aged 10 to 18 years who are clinically diagnosed with AIS and have completed a minimum of four weeks of AR-based physiotherapy delivered by licensed physiotherapists. The AR intervention incorporates visual feedback, avatar-based motion monitoring, and gamified elements to support postural correction and therapeutic engagement. Data will be collected through face-to-face, semi-structured interviews using an interview guide informed by existing literature and expert consultation. Interviews will explore how participants perceive their postural awareness, exercise motivation, adherence challenges, and psychosocial adjustments within the AR-supported environment. All interviews will be audio-recorded and transcribed verbatim. Collected data will be analyzed using Braun and Clarke's thematic analysis framework, supported by NVivo software. Two independent researchers will code the transcripts to ensure analytical rigor and thematic validity. The study is expected to contribute to the refinement of conservative scoliosis rehabilitation practices by integrating adolescent perspectives and addressing the biopsychosocial dimensions of care enhanced through technology.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 18 years
* Diagnosed with adolescent idiopathic scoliosis (AIS)
* Completed at least 4 weeks of AR-based physiotherapy
* Sufficient Turkish language proficiency to participate in interviews
* Provided written informed consent (adolescent and guardian)

Exclusion Criteria:

* Presence of neurological or cognitive conditions interfering with communication
* Withdrew before completing the intervention program
* Declined audio recording of interviews

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Awareness Following AR-Supported Physiotherapy | Within 1 week after completing the 4-week intervention
  This outcome will assess adolescents' subjective body awareness, including their perception of postural alignment, movement control, and physical self-understanding, after completing AR-supported scoliosis-specific physiotherapy. Data will be collected through semi-structured interviews and analyzed thematically to evaluate perceived changes in awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a qualitative study that involves in-depth interviews with adolescent participants diagnosed with idiopathic scoliosis. Due to the sensitive and identifiable nature of the data, individual participant data (IPD) will not be shared in order to protect confidentiality and adhere to ethical standards approved by the institutional review board. The collected data are not anonymized in a manner that would allow public sharing without risk of identification.

REFERENCES:
- [Result] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- See also: Related Info — https://scoliosisjournal.biomedcentral.com/articles/10.1186/s13013-017-0145-8